## "The effects of Neurodevelopmental Therapy on Feeding and Swallowing Activities in Children with Cerebral Palsy" NCT04403113

03.12.2019

## **Statistical Analysis Plan**

Descriptive statistics for continuous variables are expressed as mean, standard deviation values (Height, weight, body mass index (BMI), gender, etc); it is expressed as number (n) and percentage (%) for categorical variables.

In calculations, statistical significance level ( $\alpha$ ) was taken as 5% and values with P < 0.05 expressed statistical significance. "Statistical Package for Social Sciences" (SPSS 16) statistical program was used in the analysis of the data.

In statistical analysis, the suitability of all the data to normal distribution was analyzed with "One-Sample Kolmogorov-Smirnov Test" and non-parametric tests were used since the variables were not normally distributed. Chi-square test was used in binary analyzes (CP subtypes). Mann-Whitney U was used for comparing the group's data. In inter-group comparisons, the Mann-Whitney U test (pre-treatment TIS parameters and post-treatment TIS parameters; PedsQL) were analyzed. Wilcoxon test was used for intra-group comparisons.

Spearman Correlation test analysis method was used in non-parametric correlation analysis (TIS subscales and SOMA's cups, puree, semi-solids, solids and crackers after treatment).